CLINICAL TRIAL: NCT04352530
Title: Culturally Appropriate Nutrition Communication for Mexican American Women: A Randomized Controlled Trial
Brief Title: Culturally Appropriate Nutrition Communication for Mexican American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, A. Susana Ramirez, Associate Professor, University of California, Merced
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01CA190659 (NIH); K01CA190659 (NIH)
Record Dates: First submitted 2020-03-25; First posted 2020-04-20 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lifestyle Risk Reduction; Nutrition Poor; Chronic Disease; Obesity; Cancer, Breast
Keywords: sugar sweetened beverages; Health Communication; Values-based messages; Latinas; Latinx; Hispanic; Experiment; Message testing; tailoring
MeSH Terms: conditions — Risk Reduction Behavior; Malnutrition; Chronic Disease; Obesity; Breast Neoplasms | interventions — Health Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Rewind the Future (Active Comparator): Fear appeal, video message to reduce sugar consumption or risk death
  Interventions: Other: Health Communication
- Hear No (Experimental): Video of spoken word poem from The Bigger Picture project, "Hear No" by Joshua Merchant; images of African-American male poet interspersed with images of environment
  Interventions: Other: Health Communication
- The Longest Mile (Experimental): Video of spoken word poem from The Bigger Picture Project, "The Longest Mile" by Tassiana Willis; images of African-American female poet interspersed with images of environment
  Interventions: Other: Health Communication
- A Taste of Home (Experimental): Video of spoken word poem from The Bigger Picture Project, "A Taste of Home" by Monica Mendoza; images of Hispanic female poet interspersed with images of environment
  Interventions: Other: Health Communication
- Lost in Translation (Experimental): Video of spoken word poem from The Bigger Picture Project, "Lost in Translation" by Yosimar Reyes; images of Hispanic male poet interspersed with images of environment
  Interventions: Other: Health Communication
- Bottled Up (Experimental): Video of spoken word poem from The Bigger Picture Project, "Bottled Up" by Eileen Torrez; images of Hispanic female poet interspersed with images of environment
  Interventions: Other: Health Communication
- The Corner (Experimental): Video of spoken word poem from The Bigger Picture Project, "The Corner" by Jose Vadi; images of Hispanic male poet interspersed with images of environment
  Interventions: Other: Health Communication
- Thin Line (Experimental): Video of spoken word poem from The Bigger Picture Project, "Thin Line" by Ivori Holson; images of African-American female poet interspersed with images of environment
  Interventions: Other: Health Communication

INTERVENTIONS:
Other: Health Communication — Spoken word poems set to images performed by youth who wrote the poems. Videos were produced by The Bigger Project and were posted publicly to the Bigger Picture Project website and YouTube. Duration of videos ranges from 2 minutes to 6 minutes.

SUMMARY:
A randomized controlled trial to test the effects of culturally appropriate nutrition communication for Mexican American women.

DETAILED DESCRIPTION:
An unbalanced randomized controlled trial with pre-test and immediate post-test was employed to test the effects of different types of message features and appeals. The study was conducted online with Mexican American women aged 18-29 years old. Messages focused on sugary beverage consumption and the main outcomes were acceptance and receptivity to the message (i.e., perceived effectiveness), perceptions of social norms, and knowledge. The investigators also measured a number of hypothesized mediators and moderators of the effects.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latina/x or Hispanic
* Self-identify as a woman
* Self-reported as being of age between 18-29 years
* Undergraduate students enrolled in SONA at UC Merced

Exclusion Criteria:

- Not Mexican American

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self-identify as female
Enrollment: 881 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Perceived effectiveness | Immediately post-intervention
  Perceived effectiveness of the message is known to affect intention to engage in a given health behavior. Therefore, perceived effectiveness of the stimuli was assessed as a proxy measure for intention to reduce sugary beverage consumption using a 5-point, 13-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1. This scale comprised 3 subscales namely (1) Message Acceptance - 2 items, (2) Argument Strength - 4 items, (3) Personalized Perceived Effectiveness - 7 items. Greater scores on this scale represented greater levels of perceived effectiveness of the message.

SECONDARY OUTCOMES:
Identification with the message | Immediately post-intervention
  responses ranging from Strongly Agree=5 to Strongly Disagree=1. Two sample items from the scale are, "During viewing, I felt I could really get inside the person's head", and "At key moments in the video, I felt I knew exactly what they were going through". Greater scores on this scale represent greater degree of identification with the character in the video.
Activation of social justice values | Immediately post-intervention
  Activation of social justice values was measured using a 5-point, 2-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1. The two items are, "The message made me think that when I choose to eat healthy, I'm helping to make the world a better place" and "The message made me think that when I eat healthy, I'm doing my part to protect people who are being manipulated by sugary beverage companies". Greater scores on this scale represent greater levels of activation of social justice values.
Sugary beverage related media literacy | Pre-test and Immediately post-intervention
  Sugary beverage related media literacy was measured using a 5-point, 8-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1. This scale measured how much the participants understood the ways in which sugary beverage industry used media to influence and manipulate their sugary beverage consumption behaviors. Some sample items are as follows: "Certain sugary drink brands are designed to appeal to people like me", "Sugary drink ads show a healthy lifestyle to make people forget about the health risks, such as weight gain and diabetes" and "Sugary drink ads link drinking these beverages to things people want, like love, good looks, and power". Greater scores on this scale represent greater levels of sugary beverage media literacy.
Public health literacy | Pre-test and Immediately post-intervention
  Public health literacy is defined here as an understanding of the social determinants of health. This was measured using a 5-point and 7-item Likert scale with responses ranging from Strongly Agree=5 to Strongly Disagree=1. The seven items measured opinions about how much different external factors affect health because these best reflected an understanding of the social determinants of health: (1) money, (2) education, (3) safe and affordable housing, (4) early childhood experiences, and (5) government policies and programs (6) lifestyle choices and (7) consequences of system failure on the under-resourced. Greater scores on this scale represented greater levels of public health literacy.
Empowerment | Pre-test and Immediately post-intervention
  Empowerment to engage in civic action was measured using a two-item index that assessed the perceived effectiveness of engaging in civic actions. Each question was a 4-point Likert item with responses ranging from "Very Effective=4" to "Very Ineffective=1". The two items were as follows, "How effective would it be to boycott sugary beverages as a way to convince corporations to stop pushing sugar to my community?" and "How effective would it be to use social media to convince corporations to stop pushing sugar to vulnerable groups?". Greater scores on this index represented greater levels of efficacy to engage in civic action.
Beverage knowledge | Pre-test and Immediately post-intervention
  Knowledge increases self-efficacy and empowers people to make better health choices for themselves and knowledge of the negative consequences of a given health behavior increases the intention to reduce that behavior. Therefore, better knowledge of the negative consequences of sugary beverage consumption directly impacts both individual level sugary beverage consumption as well as social level psychological empowerment to advocate for reduction in sugary beverage consumption at the community level. A sugary beverage knowledge scale comprised 6 true or false items adapted from multiple studies. The statements were as follows: Excessive sugar consumption causes, (1) health problems (2) weight gain (3) dental caries (4) diabetes (5) cancer and (6) heart disease". Greater scores on this scale represented greater levels of sugary beverage knowledge.
Engagement | Immediately post-intervention
  Engagement with the message was assessed with 2 items from the Narrative Transportation Scale (Green et al.).
Similarity | Immediately post-intervention
  Perceived similarity of the participant with the main character (poet/speaker) in the video was assessed with a 2-item scale adapted from Cohen and colleagues (2018).
Elaboration | Immediately post-intervention
  Elaboration of the message arguments was assessed using a 4-point scale created by Kahlor and colleagues (2003) and a 3-point sugar-specific elaboration scale created by Dixon and colleagues (2015).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Merced SONA System (Online Platform), Merced, California, United States

IPD SHARING:
Plan to Share IPD: No